CLINICAL TRIAL: NCT06334419
Title: Placebo-Controlled, Single-Dose Challenge Study of Gaboxadol in Adult Males With Fragile X Syndrome (FXS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Craig Erickson (Other)
Collaborators: Healx Limited (Industry)
Responsible Party: Sponsor-Investigator, Craig Erickson, Research Director and Research Endowed Professor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0795
Record Dates: First submitted 2024-03-08; First posted 2024-03-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X; Fragile X Syndrome; FXS
MeSH Terms: conditions — Fragile X Syndrome | interventions — gaboxadol

STUDY DESIGN:
Intervention Model Description: This study was designed as a 2-intervention crossover, with all study participants receiving all possible interventions. These are placebo and Gaboxadol.
Masking Description: Quadruple masking (participant, care provider, investigator and outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Experimental): Participants received, in random order, a single dose of placebo or Gaboxadol with a two-week washout period between doses. The gaboxadol dosage selected for this study is 10 mg or Placebo as a single dose on each study visit (two at home and two in clinic).
  Interventions: Drug: Gaboxadol; Drug: Placebo

INTERVENTIONS:
Drug: Gaboxadol — Drug: Gaboxadol 10 mg as a single dose (two 5mg capsules)
Drug: Placebo — Two placebo capsules

SUMMARY:
This is a single dose, placebo-controlled study. Male subjects aged 18 to 40 years (inclusive) with a diagnosis of FXS. Eligible subjects may enroll in this study comprised of two in home and two in clinic visits each 14 days apart, for a total of four visits. Subjects will be given single dose gaboxadol (10 mg) or matched placebo at each of these visits to take orally. Thus, all enrolled subjects will receive placebo at home and in clinic and receive gaboxadol at home and in clinic in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject consents to participate, or if they are not their own legal guardian, offers assent supported by legally authorized representative consent
2. Subject is willing and able to comply with the study procedures as specified in the protocol and to comply with the study drug administration. Caregiver also commits to the study requirements prior to any study-related procedures
3. Subject and caregiver are both able to understand the spoken national language clearly and caregiver can read and write to complete study assessments
4. Males age 18 to 40 years (inclusive)
5. Has FXS with molecular genetic confirmation of the full FMR1 mutation (>200 cysteine-guanine-guanine [CGG] repeats). May have been confirmed historically or at Screening
6. Is in general good health as deemed by the Investigator, determined by physical examination, medical history, and laboratory tests
7. If receiving serotonin-selective reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitor (SNRI), or serotonin antagonist and reuptake inhibitor (SARI), is on a stable, well-tolerated dose for the previous 3 months with no further changes anticipated
8. Is not sexually active or can confirm at least one form of contraceptive

Exclusion Criteria:

1. Any chronic major medical comorbid condition deemed by the Investigator as presenting added risk to the subject, including but not limited to, refractory hypertension, kidney disease, or liver disease
2. Diagnosed with diabetes (Type 1 or II) or receiving any anti-diabetic medication
3. Unstable seizure disorder, defined by any seizure within 6 months prior to baseline visit and/or a change in any anti-convulsant drug dosing in the 60 days prior to study consent
4. Changes in psychotropic or anti-convulsant (where taken for reasons other than seizure control) drug treatment within 30 days prior to Screening
5. Significant changes in any educational, behavioral, and/or dietary interventions the month prior to Screening
6. Planned initiation of new, or modification of ongoing, interventions during the study
7. Unable or unwilling to take oral medication (whole capsule, despite assistance with a spoonful of applesauce, yoghurt, or equivalent liquid food)
8. Consumption of liver enzyme inducers or inhibitors including and not limited to foods, medicines, herbal remedies and supplements three days prior to any Visit. Foods or beverages containing CYP3A4/5 inhibitors (e.g., grapefruit, pomegranate, pomelo, and star fruit) should be avoided before taking study medication and for up to 1 hour post dose throughout the study
9. Has abnormal baseline laboratory assessments including, but not limited to, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin >1.5 × the upper limit of normal (ULN), serum creatinine >1.5 x ULN or other clinically relevant laboratory abnormality
10. Has a clinically significant heart rate or blood pressure (BP) at Screening as judged by the Investigator
11. Has received an investigational drug in any prior clinical study within 30 days or 5 half-lives (whichever is longer) prior to Screening

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
To evaluate target engagement of gaboxadol treatment on high density EEG recordings | Pre-dose, 60 minutes post-dose
  Changes in EEG recordings with gaboxadol treatment (60-90 minutes post-dose compared with pre-dose on resting theta, alpha and gamma band relative and absolute power; brain response to auditory chirp stimuli in the gamma band range).

SECONDARY OUTCOMES:
To investigate the feasibility of home research visits and procedures in adult males with FXS | Pre-dose, 60 minutes post-dose
  Quality and test-retest reliability of assessments performed at home compared with the hospital setting. This includes blood testing for Fragile X messenger ribonucleoprotein (FMRP: range of 0-40 picomolar) and eye-tracking of eye gaze to eye regions when viewing faces (range of value from 0 percent to 100 percent; higher values are associated with a neurotypical phenotype).
To investigate the feasibility of high density EEG recording at home in adult males with FXS | Pre-dose, 60 minutes post-dose
  Quality of EEG recordings in the home setting compared with EEG recordings performed in the hospital setting. We will compare the duration of usable artifact free EEG resting data from the same subject gathered at home and at clinic.
To potentially explore the pharmacokinetics of gaboxadol treatment in single-dose trial design | Pre-dose, 60 minutes post-dose
  PK profile (the level of gaboxadol in human plasma) will be obtained at 60 +/- 10 minutes post-dose only).
To investigate the effect of gaboxadol treatment on neuropsychological assessments | Pre-dose, 60 minutes post-dose
  Changes in cognitive and neuropsychological assessment measures with gaboxadol treatment (RBANS). RBANS list learning subscale score range is -4 to +4, higher values are indicative of greater memory.
To investigate the effect of gaboxadol treatment on eye tracking assessments | Pre-dose, 60 minutes post-dose
  Change in eye tracking outcomes (60-90 minutes post-dose compared to pre-dose on percent viewing of social versus geometric scene
To investigate the effect of gaboxadol treatment on clinician-rated measures | Pre-dose and post-dose
  Change in clinician-rates measures (post-dose compared to pre-dose on CGI-I)
To determine whether FMRP levels predict treatment response | Pre-dose and post-dose
  Relationship between FMRP (Fragile X messenger ribonucleoprotein) level and degree of change (baseline/screen to post-dose) across measures

CONTACTS AND LOCATIONS:
Overall Officials: Cragi A Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States